CLINICAL TRIAL: NCT04103827
Title: Usability Assessment of a Device to Promote Physical Activity for Old Patients Hospitalized
Brief Title: Qoos Use Sustaining Health Among patIents hOspitalized in Geriatric mediciNe (QUSHION)
Acronym: QUSHION
Status: Withdrawn | Type: Observational
Why Stopped: no patient included after 6 month of enrollement
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019/40
Record Dates: First submitted 2019-09-13; First posted 2019-09-25 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Old Age; Usability; Satisfaction
Keywords: Usability; Elderly; Old people; Physical activity; Balance
MeSH Terms: conditions — Personal Satisfaction; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- old patients: During the first 24 hours of the hospitalisation in the equiped room and before the presentation of the device, A first series of questions will be asked a priori to the patients. Patient will freely use "Le Qoos" during all his hospitalisation. After this use, a survey concerning the usability of "Le Qoos" will be administered to the patient, during the 48 hours before his discharge from hospital.
  Interventions: Other: usability assessment
- relatives / unformal caregivers: Before the presentation of the device, a first series of questions will be asked a priori to the unformal caregiver. Unformal caregiver will freely use "Le Qoos" during the hospitalization of his relative. After this use, a survey concerning the usability of "Le Qoos" will be administered to the unformal caregivers, 48 hours before the discharge of his hospitalized relative from hospital.
  Interventions: Other: usability assessment
- profesional caregivers: After the inclusion of all expected patients and relatives, a survey concerning the usability of "Le Qoos" will be administered to professional caregivers.
  Interventions: Other: usability assessment

INTERVENTIONS:
Other: usability assessment — Usability of "Le Qoos" will be assessed using a validated usability questionnaire

SUMMARY:
Falls are a frequent and serious problem in old people. It is estimated that one-third of subjects over 65 years of age and 50% of those over 85 years of age have at least one fall per year (1). The traumatic and psychological consequences of falls contribute to the loss of functional independence and lead to early institutionalization (2).

All activities of daily living require us to maintain a state of postural balance, whether standing, sitting, static or dynamic. Thus, good coordination is essential to maintain balance, reflecting both peripheral (muscular) and central (cognitive) motor control (3,4). Coordination skills between posture and movement decline during aging without associated disorder, and even more so when this aging is associated by cognitive disorders (5,6).

On the contrary, as part of a balance rehabilitation program, an adapted training allows the partial recovery of the balance management process in elderly subjects who fall (7).

Le Qoos® by LudHealth is technical foam equipment, which can be installed on the wall, to practice various physical exercises. It can therefore be used as a simple support, leaning on with hands, arms, feet or even the head, exerting contact points, pressures or even impacts with more or less force. Le Qoos® is an equipment that allows to perform, on the same object, gentle or tonic exercises, balance, flexibility, sheathing or muscle strengthening while having fun.

We hypothesize that cognitive-physical stimulation workshops based on the use of the device Le Qoos® and is environment are i) adapted to geriatric fall prevention issues, ii) accessible to elderly hospitalized patients and health professionals, and iii) effective and safe to maintain and/or recover postural balance in elderly hospitalized patients.

First step of this work is to assess whether "Le Qoos" is considered as usable par end-users of the device.

DETAILED DESCRIPTION:
This satisfaction survey will be carried out in the Geriatrics department of the University Hospital of Angers. Actually, Le Qoos and is environment is installed in a hospitalisation room of the geriatric unit. When the patient entered the room, a first series of questions are asked a priori concerning the device. These questions are also asked to the relatives of the patient if any, and to the professional caregivers of the unit. After this first series of questions, a list of possible exercises is given to the patients, regrading is functional capabilities according to the EGS-1, with some explanations. The proposed exercises correspond to 3 selected actions based on the results of scientific research conducted by the team at the University Hospital of Angers to prevent the risks of iatrogenic dependence. Then, the patient and is relatives, if any, are free to use the device during the all hospitalisation. During the 48h before the discharge from the hospital, a second list of questions will be asked to assess the usability and the satisfaction concerning the device.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Aged 65 years old and over
  * To be hospitalised in geriatric medicine department of Angers University Hospital
* Caregivers:

  * Family members or relatives
  * Aged 18 years old and over
* Healthcare team :

  * geriatric medicine department's staff of Angers University Hospital
  * Aged 18 years old and over

Exclusion Criteria:

* To be under legal protection
* Refusal of participating

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients are recruited during their hospitalisation in geriatric medicine. Relatives / unformal caregivers are recruited during the hospitalisation of patients in geriatric medicine.
  Professionnal caregivers are recruited in the acute care geriatric unit.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-09-16 (Estimated); Study Completion 2020-10-05 (Estimated)

PRIMARY OUTCOMES:
Usability of the device "Le Qoos" | During the 48 hours before the discharge of the hospital
  The usability will be assessed using the validated System Usability Scale (SUS). SUS scale range from 0 to 100. The mean score obtained by users will be calculated. A score over 50 could be considered as acceptable usability. A score over 65 could be considered as good usability.

SECONDARY OUTCOMES:
Satisfaction of the users following the use of the device "Le Qoos" | During the 48 hours before the discharge of the hospital
  The satisfaction will be assessed using a non-validated satisfaction questionnaire based on a forced choice Likert scale in 4 points from 1 to 4. The mean score obtained by users will be used. Users will be considered as satisfied if the mean score is over 2 on 4.
Frequency of use of the device "Le Qoos" by elderly hospitalized patients. | During the 48 hours before the discharge of the hospital
  The frequency of use will be described using a non-validated questionnary based on 4 closed questions.
The most appreciated ergonomic elements | During the 48 hours before the discharge of the hospital
  The ergonomic elements will be assessed using a single choice closed liste of ergonomic elements. The most ergonomic elements will be ranked in descending order of citation by users.
Areas of improvment regarding ergonomics of "Le Qoos" | During the 48 hours before the discharge of the hospital
  A single open question will be asked for users concerning elements to improve. A qualitative thematic analyze of the verbatim will be realized to identify the elements to improve,

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Annweiler, MD, PhD, Principal Investigator — Angers University Hospital
Locations (1):
- Angers University Hospital, Angers, France